CLINICAL TRIAL: NCT02567864
Title: Development and Evaluation of an Evidence-based Intervention Guideline of the Healthy Beat Accupunch (HBA) Exercise Program for the Community Older Adults
Brief Title: Development and Evaluation of the Healthy Beat Accupunch (HBA) Exercise Program for the Community Older Adults
Acronym: HBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUH-IRB-20140089
Record Dates: First submitted 2015-09-29; First posted 2015-10-05 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Functional Fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Beat Accupunch (Experimental): The HBA exercise program includes: 1) warm-up: 5 slow and gentle exercises to regulate qi, loosen up the body, and elevate the energy for a safe transition to the next phase, 2) accupunch: 14 low-to-medium speed exercises to punch the 14 meridians to enhance the cardiovascular-respiratory workout, and 3) relaxation: 5 low-speed, muscle relaxing exercises with deep breaths to sooth the body and mind. It is conducted 3 times per week and 40 minutes per practice.
  Interventions: Other: Healthy Beat Accupunch exercise program
- control (Active Comparator): The control group maintains daily activities.
  Interventions: Other: control

INTERVENTIONS:
Other: Healthy Beat Accupunch exercise program — HBA has three phases and takes 40 minutes to complete.
  Arms: Healthy Beat Accupunch
Other: control — participants maintain their daily activities.
  Arms: control

SUMMARY:
The goals of this research project were: 1) to develop a senior-tailored Healthy Beat Accupunch (HBA) exercise program for community-dwelling older adults, 2) to test the effects of a six-month, instructor-led HBA exercise program, and 3) to evaluate the feasibility, compliance, and long-term effects of a six-month, DVD-guide HBA exercise program.

DETAILED DESCRIPTION:
A three-year, longitudinal, triangulation research method was applied. First Year (Phase I): A preliminary HBA exercise program, including hard copy descriptions and DVD demonstrations of each exercise, was mailed to the 16 experts in the Delphi advisory panel for their critique and evaluation. First Year (Phase II): A quasi-experimental, one-group, pretest-posttest design was used to pilot-test the feasibility of the HBA exercise program on a group of 31 community-dwelling older adults in a community care station. Second Year: A cluster randomized controlled trial was used to test the effects of a six-month, instructor-led HBA exercise program on the functional fitness (cardiovascular-respiratory function, body flexibility, muscle strength, and muscle endurance) of the community-dwelling older adults. Through the use of convenience sampling strategy, eight community care stations with 232 older adults in Kaohsiung were recruited and randomly assigned based on their community care stations to a HBA experimental group or a wait-list control group. Participants in the experimental group received the HBA exercise program led by trained and certified instructors, three times per week, 40 minutes per practice for six months; participants in the wait-list control group continued with their regular daily activities. One pre-test and two post-tests, three months apart, were conducted. Third Year: Using the same method as in the second year, participants from the second year continued practicing the HBA exercise program, but guided by a DVD, for another six months. The feasibility, compliance, and effectiveness of the DVD-led HBA exercise program on the community-dwelling older adults were tested, and another two post-tests, three months apart, were conducted on the same outcome measurements as in the second year.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older adults aged 65 and over
* Mandarin or Taiwanese speakers
* able to stand and walk without assistive devices
* cognitive alert and able to verbally state their name, address, and answer questions.

Exclusion Criteria:

* participants with severe and acute cardiovascular, musculoskeletal, or pulmonary illnesses.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-07-12 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Digital Sphygmomanometer | 12 months
  Blood Pressure
TruZoneTM Peak Flow Meter | 12 months
  Lung Capacity
Two-minute Step Test | 12 months
  Aerobic Endurance
Back Scratch Test | 12 months
  Upper Body Flexibility
Chair Sit-and-Reach Test | 12 months
  Lower Body Flexibility
Digital Handgrip Dynamometer | 12 months
  Hand-Grip Strength
Arm Curl Test | 12 months
  Upper Limbs Muscle Endurance
Chair Sit-to-Stand Test | 12 months
  Lower Limbs Muscle Endurance

SECONDARY OUTCOMES:
Barthel Index | 12 months
  ADL
chronic pain | 12 months
  pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan